CLINICAL TRIAL: NCT06655402
Title: Efficacy and Sustainability of a Carepartner-Integrated Telerehabilitation Program for Persons With Stroke
Acronym: CARE-CITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sarah Blanton, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00007645; R01HD115644 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Caregiver Burden
Keywords: Stroke Survivors; Carepartners; Caregivers; Post-Stroke Recovery; Telehealth; Rehabilitation
MeSH Terms: conditions — Stroke; Caregiver Burden | interventions — Control Groups; Accelerometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CARE-CITE- CarePartners (Intervention Group) (Experimental): The CP will receive virtual Collaborative Integrated Therapy (CARE-CITE), a post-stroke family education program.
  Interventions: Behavioral: CARE-CITE
- CARE-CITE- Stroke Survivors (Intervention Group) (Experimental): This study arm consists of stroke survivors (SS) of carepartners receiving the virtual Collaborative Integrated Therapy (CARE-CITE), a post-stroke family education program.
  Interventions: Behavioral: CARE-CITE; Other: Actigraph GT3X+
- Attention Control Group-CarePartners (Active Comparator): CP in this group will receive traditional written family educational materials to review during the 4-week intervention period.
  Interventions: Behavioral: Attention Control Group
- Attention Control Group-Stroke Survivors (Active Comparator): This study arm consists of stroke survivors (SS) of carepartners receiving the traditional written family educational materials to review during the 4-week intervention period.
  Interventions: Behavioral: Attention Control Group; Other: Actigraph GT3X+

INTERVENTIONS:
Behavioral: CARE-CITE — CARE-CITE is a post-stroke family education program, to support care partners (CPs) in aiding stroke survivors (SS) during rehabilitation. Utilizing autonomy-supportive strategies, CARE-CITE emphasizes empathy, choice, and problem-solving while minimizing controlling language.
  The program features a user-friendly web-based platform with interactive videos that guide CPs in providing support for SS. Over four weeks, CPs engage in two virtual home visits and two phone check-ins. During the initial visit, CPs review online modules, set collaborative goals, and co-create a home exercise plan targeting upper extremity (UE) activities. The second and third weeks involve structured phone calls to discuss autonomy-supportive strategies and address challenges.
  The final visit reinforces strategies, assesses SS progress, and adjusts rehabilitation goals. Each module is designed to foster motivation and effective practice in daily activities.
  Other Names: Carepartner and Collaborative Integrated Therapy
  Arms: CARE-CITE- CarePartners (Intervention Group); CARE-CITE- Stroke Survivors (Intervention Group)
Behavioral: Attention Control Group — Over a similar 4-week period, the SS and CP will receive the same number of structured virtual weekly visits as the CARE-CITE group without the review of CARE-CITE modules.
  The CP will receive a brochure with general caregiving information and website resources. At week 1, a separate control group intervention therapist will deliver a 2-hour virtual home visit to evaluate SS UE function and assess safety concerns. Based on SS impairments, a home exercise program will be prescribed for flexibility, strength, and coordination (6-8 exercises, 2 sets of 10 reps). SS will be encouraged to practice daily (targeting 30 min/day). Weeks 2 and 3: CP Phone check-ins [15-minute]. The intervention therapist will review safety, assess adverse events, and CP's use of web resources. Week 4 Virtual Home visit (2 hours). Review SS's progress with the UE activity home exercise program, discuss safety concerns, and progress UE exercises as appropriate.
  Other Names: Control Group
  Arms: Attention Control Group-CarePartners; Attention Control Group-Stroke Survivors
Other: Actigraph GT3X+ — Accelerometry data will be collected using Actigraph GT3X+ wearable sensors, approved by the FDA. The device does not collect or store individually identifiable health information (IIHI), private health information (PHI), or sensitive data. It is not intended for diagnosing, treating, or preventing diseases. These small, wrist-worn monitors document physical movement for physiological monitoring, including tracking movement during sleep. They can analyze circadian rhythms and assess activity in situations where quantifiable analysis of physical motion is needed.
  Other Names: Accelerometry
  Arms: Attention Control Group-Stroke Survivors; CARE-CITE- Stroke Survivors (Intervention Group)

SUMMARY:
Stroke is a leading cause of long-term disability. Research has placed little emphasis on integrating care partners (CP) (family members) into the rehabilitation process without increasing negative care partner outcomes. The research team has developed and implemented a novel, web-based care partner-focused intervention (CARE-CITE) designed to foster problem-solving and skill building while facilitating care partner engagement during stroke survivor (SS) upper extremity practice of daily activities in the home setting. By providing a family-focused approach to rehabilitation interventions, this project will help develop more effective treatments that improve CP and outcomes after stroke.

DETAILED DESCRIPTION:
The goals of this study are to use a fully virtual, two-group randomized clinical trial to assess the efficacy of CARE-CITE and the sustainability of improvements compared to an attention control group.

The specific aims are to determine the effects of CARE-CITE on stroke survivors' upper extremity functional capacity (Aim 1), upper extremity daily activity performance (accelerometry and patient-reported measures), and social participation (Aim 2). Additionally, the investigators will evaluate the effects on care partner strain, conflict around stroke recovery, and quality of life (Aim 3).

Study participants will be identified and recruited within the Emory Healthcare system and regional Atlanta hospitals, partnering with clinical staff for referrals and meeting with local stroke support groups. All Emory Rehabilitation Hospital stroke admissions will be screened based on study inclusion/exclusion criteria and contacted by the research coordinator, if eligible. The project coordinator will make a virtual screening appointment for interested participants. If screening criteria are met, the informed consent will be reviewed and obtained virtually to enroll the dyad.

Individual participant's enrollment in the study will last 29 weeks. All study visits will be virtual. Over 4 study evaluation sessions (~2hrs/dyad), the research team will collect stroke survivor (SS) and care partner (CP) data at baseline and after the intervention using questionnaires and objective measures of upper extremity recovery. Upper extremity recovery will be evaluated by direct observation during the virtual assessments and through wearable sensors (worn on the stroke survivor's wrists for 3-7 days during the assessment periods).

The intervention will last 4 weeks. During the intervention period, dyads in both the intervention and attention control groups will receive two virtual home visits and two phone check-in visits. A research therapist will guide the SS and CP in the development of goals and a home exercise program to improve the upper extremity function of the SS. During the follow-up period, dyads will receive one 30-minute check-in booster call and a 2-hour booster virtual home visit. Care Partners in the intervention group will review CARE-CITE during the 4-week intervention period. CARE-CITE is a user-friendly, web-based program that features exemplary and interactive videos of family scenarios surrounding upper extremity rehabilitation at home. CP in the Attention Control group will receive traditional written family educational materials to review during the 4-week intervention period.

Aligned with the NIH Research Plan on Rehabilitation, this work will impact the development of innovative family-level interventions to improve SS and CP outcomes.

ELIGIBILITY:
CarePartners (CP):

Inclusion Criteria:

* Must be at least18 years old,
* Able to read and write English,
* Mini-mental test score greater than 24
* Individuals who are a spouse/partner or family member dwelling in the same household and self-identify as the primary caregiver of the SS.

Stroke Survivors (SS):

Inclusion Criteria:

* Must be at least18 years old
* More than 3 months and less than 2yrs post-ischemic or hemorrhagic event
* Discharged home from the hospital with minimal to moderate UE deficits (can actively initiate 20 degrees of wrist and 10 degrees of finger extension)
* Mini-mental test greater than 24
* No physician determined medical problems that would limit participation,
* Must have CP living in the home

Exclusion Criteria for CP and SS:

* Significant cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
SS's Upper Extremity Functional Capacity | Baseline, 2 months and 6 months post-intervention
  Upper Extremity Fugl Meyer (FM) therapist standardized assessment. Total score=sum of 33 items; range 0-66 higher score, less UE impairment.
SS's UE activity performance using the Motor Activity Log (MAL) | Baseline, 2 months and 6 months post-intervention
  MAL, a 30-item questionnaire, Likert-type scale, assessing the use of the affected arm during normal daily activities. Responses are given on a Likert-type scale where 0= the weaker arm was not used at all for that activity (never) to 5=the ability to use the weaker arm for that activity was as good as before the stroke (normal). The total scores are the average of all items and range from 0 to 5, where higher values indicate the greater function of the arm impacted by the stroke. A high score/high-quality UE use.
SS's Social Participation Score using the Stroke Impact Scale (SIS) score | Baseline, 2 months and 6 months post-intervention
  Stroke Impact Scale (SIS), is a stroke-specific self-report questionnaire (59 items across 8 domains) that measures how a stroke has impacted a participant's health. The Social Participation Domain: rated in a 5-point Likert scale regarding the difficulty the participant has experienced completing each item (range 0-100). Higher scores, higher social participation.
CP Quality of Life | Baseline, 2 months and 6 months post-intervention
  CP will complete the Bakas Caregiving Outcomes Scale (BCOS). BCOS is a unidimensional scale based on 15 items and addresses changes in caregiving social functioning, subjective well-being, and physical health. Participants respond to statements on a 7-point Likert scale (-3 =changed for the worst, +3 = changed for the best, with 0 meaning did not change). The -3 to +3 ratings are recoded to 1-7 so positive numbers used for analysis. Total BCOS score ranges from 15-105. A Cut-off score >60 = positive life changes. Higher scores, better caregiving outcomes.
CP Strain using the Caregiver Strain Index(CSI) | Baseline, 2 months and 6 months post-intervention
  Caregiver Strain Index (CSI), self-reported. A 13-question tool that measures strain related to care provision with binary yes/no answers. There is at least one item for each major domain: Employment, Financial, Physical, Social, and Time. Scoring ranges from 0 to 13, with scores of 7 or more indicating a greater level of stress. Higher scores, more strain.

SECONDARY OUTCOMES:
SS Upper Extremity Functional capacity (ArmCAM) | Baseline, 2 months and 6 months post-intervention
  Arm Capacity and Movement Test (ArmCAM). A therapist standardized assessment. A 10-item scale (range = 0-30); designed specifically to evaluate UE motor function virtually by videoconferencing.
SS's Upper Extremity activity performance (accelerometry) | Baseline, 2 months and 6 months post-intervention
  Accelerometers will be worn for all activities over 3-7 days except for water-based activities. These activities include activities of daily living. Accelerometry data will be gathered via Actigraph GT3X+ wearable sensors per FDA definition and approval of device use. After the virtual baseline (T0) data collection visit, the blinded data collector (licensed physical or occupational therapist) will review the accelerometer procedures with the dyad, confirm proper donning and UE wrist placement of the devices, and wear-time of 3-7 days.
Family Conflict using the Family Caregiver Conflict Scale (FCCS) score | Baseline, 2 months and 6 months post-intervention
  The FCCS is a unidimensional, Likert-type scale composed of 15 items. Each item response is in a Likert-type format with participants indicating their agreement with the item with 1 "not true at all" to 7 "very true." Item scores are summed and higher scores represent higher levels of conflict within a family. Total scores Range 15-105.
Autonomy Support Family Care Climate Questionnaire for Carepartner (FCCQ-CP) Scale Score | Baseline, 2 months and 6 months post-intervention
  Autonomy support for carepartners will be assessed by the Autonomy Support Family Care Climate Questionnaire for Carepartner (FCCQ-CP) Scale. An autonomy-supportive environment is characterized by empathy, communicating choices (avoiding controlling language), providing rationales and problem-solving. Questions are asked about the carepartner's perspective on how much they provide an autonomy supportive environment for the stroke survivor. The FCCQ-CP includes 14 items scored from 1 to 7 where 1 = not true at all and 7 = very true. Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the carepartner thinks they are providing high autonomy support to the stroke survivor.
Autonomy Support Family Care Climate Questionnaire for Stroke Survivor (FCCQ-SS) Score | Baseline, 2 months and 6 months post-intervention
  Autonomy support will be assessed using the Autonomy Support Family Care Climate Questionnaire for Stroke Survivors (FCCQ-SS). An autonomy-supportive environment is characterized by empathy, communicating choices (avoiding controlling language), providing rationales, and problem-solving. Questions are asked about the stroke survivor's perspective on how much the carepartner provides an autonomy-supportive environment for the stroke survivor. The FCCQ-SS includes 14 items scored from 1 to 7 where 1 = not true at all and 7 = very true. Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the stroke survivor perceives receiving high autonomy support from the carepartner.
SS UE self-efficacy using the Confidence in Hand and Movement Scale (CAHM) score | Baseline, 2 months and 6 months post-intervention
  Stroke survivor UE self-efficacy will be assessed with the CAHM Scale. The CAHM is a 20-item questionnaire where the items are scored on a scale of 0 (very uncertain) to 100 (very certain) and averaged to provide a total score ranging from 0-100; higher scores indicate greater confidence in performing daily tasks with the impacted arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Blanton, PT, DPT, Principal Investigator — Emory University
Locations (1):
- Emory Rehabilitation Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator will share de-identified participant-level data in both raw and pre-processed forms on NICHD DASH to facilitate replication and validation of findings associated with each aim.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Investigators will share data associated with a publication through DASH no later than the first date of the electronic publication and will share all study data by the end of the award performance period.
Access Criteria: The research community will have access to the data when the award ends. The data will be preserved indefinitely and is subject to decisions by NICHD DASH.
URL: https://dash.nichd.nih.gov/resource/submission